CLINICAL TRIAL: NCT06897774
Title: Does Transcutaneous Phrenic Nerve Stimulation Prevent Diaphragm Atrophy?
Acronym: NMES
Status: Recruiting | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, Safiye Tuba Kaplan, Doctor, Bakirkoy Dr. Sadi Konuk Research and Training Hospital
Other Study IDs: z2g6egpa
Record Dates: First submitted 2025-03-06; First posted 2025-03-27 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Critical Care, Intensive Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Early Group: The group in which transcutaneous electrical nerve stimulation will be inserted immediately after intubation
- Late Group: The group to be fitted with transcutaneous electrical nerve stimulation 48 hours after intubation

SUMMARY:
Dear participant Participants's patient, who is participants's first-degree relative, who is connected to a ventilator in the intensive care unit, unconscious and not authorized to give informed consent, has been invited to participate in the study titled 'Does transcutaneous phrenic nerve stimulation prevent diaphragm atrophy?

In order to strengthen this muscle and prevent loss of function, investigator provide electrical stimulation between the rib cage and abdomen through the skin with the tens device, causing the muscle to contract and enabling our patient to leave the respirator early.

Investigator aimed to investigate the protective effect of the tens device on the diaphragm by evaluating the diaphragm muscle with the ultrasonography device during the period when it is connected to the respirator. For this reason, the diaphragm will be contracted by giving electrical stimulation three times a day for 30 minutes with the tens device for 5 days during the period when participants's patient is connected to the respirator, and intermittent diaphragm ultrasound will be evaluated.

Participants or participants's legal guardian are asked to approve the use of participants's medical records during participants's treatment in the intensive care unit, provided that participants's personal information is kept confidential. Participants will not incur any financial burden by participating in the study and participants will not receive any additional payment.

Participants are free to leave the study at any time if deemed necessary, and the researcher can terminate the study if deemed necessary. The information obtained within the scope of the research can be used for scientific purposes and can be presented and published provided that the confidentiality record is respected.

I have read (or orally listened to) the text above, which contains the information given to the participants before the research began. I agree to participate in the study as a Volunteer. I consent to the use of my medical information. I also understand that if I do not agree to participate in the study, my treatment will be carried out in full without interruption.

Participant name and surname:

Participant's relative's name and surname:

Degree of closeness:

Signature / Date:

DETAILED DESCRIPTION:
In our study, investigator will investigate the effects of early and late trancutaneous phrenic nerve cytimulation on the prevention of diaphragm atrophy in invasive mechanical ventilation patients (>72 hours MV requirement).

Material and Methods of the Study Our study was planned as prospective, single-center, observational. As a result of the power analysis investigator performed for our study, the minimum sample size was calculated as 40 people for each group and 80 people in total with a 90% confidence interval.

Our study will be conducted as specified in the 1995 Declaration of Helsinki

The patients admitted to the Intensive Care Unit of the Anesthesia and Reanimation Clinic of the University of Health Sciences Bakırköy Dr. Sadi Konuk Training and Research Hospital Anesthesia and Reanimation Clinic Intensive Care Unit between February 1, 2024 and February 1, 2025, the effects of early and late transcutaneous phrenic nerve cytimulation on the diaphragm, diaphragmatic ultrasound and the patient's data registered in the Metavision /QlinICU Clinical Decision Support Software System will be obtained by Structured Query Language (SQL) queries. Vital parameters, hemodynamic, ventilator parameters, laboratory and demographic data will be extracted from the data pool.

Demographic data, biochemical parameters, comorbidities, indications for intubation, duration of invasive mechanical ventilation, respiratory rate, saturation, tidal volume, compliance, FiO2, Peep, above Peep, weaning criteria, peak heart rate, systolic & diastolic blood pressure, Mean arterial pressure, nutritional assessment, balance status, sedation status, length of ICU and hospital stay, and SOFA, APACHI II, Charlson comorbidity Index (CCI) and Ramsey sedation scores will be extracted from the electronic data system to homogenize the groups.

Patients will be divided into two groups according to early and late transcutaneous electrical diaphragmatic stimulation (TEDS). Group 1 patients with early TEDS will start TEDS at T1 and continue for 5 days. Group 2 patients receiving late TEDS will start TEDS at T2 and continue for 5 days.

Patients receiving invasive mechanical ventilation will receive transcutaneous electrical diaphragmatic stimulation (TEDS) for 30 minutes at 8-hour intervals for 5 days, starting immediately after intubation (0.hour) and 48 hours later. During each session, round electrodes will be placed in the parasternal region, near the xiphoid process, and in the sixth and seventh intercostal spaces in line with the mid-axillary line. TEDS will be performed using a commercial stimulator (Longest MStim Reha LGT_231 portable Electro-Stimulation Therapy Device/China) that applies electrical waves with a frequency of 60Hz, a pulse width of 300 μs and a strength of 30 milliamps. Each stimulation will be applied for 30 seconds: 5 seconds rise time, 5 seconds stimulation time, 5 seconds descent time, 15 seconds listening time. Each session will last 30 minutes and will be performed three times a day. 60 stimulations per session and 180 stimulations per day will be applied to the patient. Stimulation will not be applied when patients are under curare, in pron position, hemodynamically unstable despite catecholamines and agitated (Ramsay sedation score 1/6). The cycles would not be fully synchronized with inspiration as the patients would be ventilated in controlled and pressure support modes.

Patients will undergo diaphragm evaluation with ultrasonography at certain time intervals.

T1: intubation +4h T2: 48.hour+ 4h T3: day 5+4h US-guided diaphragm measurements will be performed in the semi-recumbent position. For evaluation of diaphragm thickness parameters, the diaphragm will be visualized by placing the 7 MHz transducer in the apposition zone perpendicular to the chest wall, in the eighth or ninth intercostal space, between the anterior axillary and midaxillary lines. The diaphragm will be visualized as a structure consisting of two echoic lines (diaphragmatic pleura and peritoneal membrane) and a hypoechoic structure between them (the muscle itself). During quiet tidal breathing, several images of the diaphragm will be taken, at least three at the point of inspiration and at least three at the end of expiration. In each B-mode image, the diaphragm thickness (Tdi) will be measured from the center of the pleural line to the center of the peritoneal line. These three measurements will be averaged and then the diaphragm thickness fraction (DTF) will be calculated as a percentage using the following formula: (End-inspiratory thickness - End-expiratory thickness)/ End-expiratory thickness. To assess the movement of the diaphragm, the 3.5 MHz probe will be placed in the mid-clavicular line below the right subcostal border and moved until the posterior third of the right diaphragm is better visualized. During tidal breathing, M-mode will be used to visualize diaphragm movement along a selected line perpendicular to the diaphragm.

Transcutaneous electrical diaphragm stimulation for both groups will be used in our daily practice.

Patients will be scheduled at the frequency and in the way of application that investigators routinely apply and the routine will not be deviated from.

Statistical Method

GraphPad Prism (v 5.01) program will be used for statistical analysis of the findings obtained in the study. Homogeneity of the variables will be determined by Shapiro-Wilk normality test. Pairwise comparisons of the groups' parameters and demographic data will be compared by Mann Whitney U test, and median and interquartile range (IQR) values will be used in statistical representation. Frequency distribution and percentage values of categorical variables such as gender and intensive care mortality will be compared with the Chi-square test. Within-group repeated measures will be compared by Wilcoxon test for pairwise comparisons and repeated MANOVA for multiple comparisons of more than two parameters. Benforini tests will be used to determine whether there is a statistical difference between the variances. For the statistical representation of the Repeated MANOVA method results, the difference between means and the standard deviation values of the differences will be used. Among the statistical values, p < 0.05 will be considered significant. In the power analysis performed to determine the sample size, the number of patients required to be in each group for the power of the study to be above 80% was calculated as 40. Thus, the number of patients to be included in the study for both groups was calculated as 80.

ELIGIBILITY:
Inclusion Criteria:Patients on invasive mechanical ventilation for 72 hours or more Patients older than 18 years

Exclusion Criteria: Patients under 18 years of age

* Patients with less than 72 hours of mechanical ventilation
* Pregnancy
* Patients with a body mass index above 35kg/m²
* Neuromuscular disease
* Refractory epilepsy
* Patients with pacemakers
* ARDS
* Unilateral or bilateral diaphragm paralysis
* Presence of pneumothorax
* Patients with large right pleural effusion
* Tracheostomized patients
* Patients undergoing upper abdominal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on invasive mechanical ventilation for 72 hours or more Patients older than 18 years
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-04-22 (Estimated); Study Completion 2025-04-22 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome: Diaphragm atrophy, ventilator-associated diaphragm dysfunction | January 22 2024-April 22 2025
  By performing phrenic nerve stimulation with TEDS device, the thickness change in the diaphragm muscle will be measured by usg at the end of 5 days.
  The thickness of the diaphragm muscle will be measured in inspiratory and expiratory. Atrophy will be determined according to the change in thickness. Diaphragm thickening fraction will be calculated by formilizing the thickness in inspiratory and expiratory and diaphragm dysfunction will be determined.DTF (End-inspiratory thickness - End-expiratory thickness)/ End-expiratory thickness)x100. The following values will be accepted for the results.
  Diaphragmatic Atrophy:
  Diaphragm thickness<1-1.5cm Diaphragmatic thickness decreased by 10% compared to baseline
  Diaphragmatic Dysfunction:
  Diaphragmatic Thickening Fraction <20

SECONDARY OUTCOMES:
1.Duration of Mechanical Ventilation 2.Length of Stay in Intensive Care Unit | January 22 2024-April 22 2025
  1. Definition: Total duration of mechanical ventilation received by the patient. Unit of Measure: Hours
  2. Definition: Total length of stay in the intensive care unit. Unit of Measure: Days

CONTACTS AND LOCATIONS:
Locations (1):
- Dr.SadiKonuk EAH, Istanbul, Bakirkoy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
I haven't decided yet